CLINICAL TRIAL: NCT00749164
Title: Allogeneic Mesenchymal Stem Cell Infusion for Treatment Of Steroid Resistant GVHD
Brief Title: Allogeneic Mesenchymal Stem Cell for Graft-Versus-Host Disease Treatment
Acronym: MSCGVHD
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Prof. Igor B. Resnick, Hadassah Medical Organization
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IBR-0137-08-HMO-CTIL
Record Dates: First submitted 2008-07-14; First posted 2008-09-09 (Estimated); Last update posted 2009-08-11 (Estimated); Status verified 2009-08

CONDITIONS: Graft-Versus-Host Disease
Keywords: Mesenchymal stem cells; Umbilical cord; graft-vs-host disease; Steroid resistant
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: MSC transplantation — 1-2X10^6 MSC per kg

SUMMARY:
Now it is commonly accepted that MSC produce an immune-tolerant environment in different settings. It has been shown (mainly for BM-MSC) that MSC can down-regulate T cells activation. This characteristic of BM derived MSC already has clinical implications and shows their potent effectiveness both in prophylaxis and treatment of resistant GvHD. Ongoing clinical trials of use bone marrow MSC for treatment of steroid resistant GvHD are successfully run on and some bone marrow donor registries included BM-MSC as a material for donation. According to our preclinical studies MSC from cells from marrow, placenta, umbilical cord vessels demonstrate similar pronounced immunosuppressive effect both with autologous and allogeneic lymphocytes. Our preliminary clinical experience shows that BM-MSC is an effective tool for treatment of steroid resistant GVHD. Present study aimed to demonstrate if human UC-MSC has in vivo immunosuppressive effect and can be used for GVHD treatment

ELIGIBILITY:
Inclusion criteria:

1. Informed consent. 2. Any patient that has undergone allogeneic stem cell transplantation with steroid refractory grades II-IV acute GvHD either occurring post transplant, or induced by donor lymphocyte infusions (DLI) or T-cell add back. A positive biopsy for GvHD is not required if clinical signs and symptoms are characteristic for GvHD and other etiologies are excluded.

3. Patient received best known therapy for GvHD including: i. Patients must receive cyclosporine A (trough level 150-300 ng/ml) or tacrolimus (trough level 5-15 ng/ml).

ii. In addition, steroids must have been given, for instance prednisolone ≥2 mg/kg/day (or equivalent doses of methylprednisolone, etc.) for at least 72h in case of progressive acute GvHD, 5 days non progressive acute GvHD.

iii. Despite this treatment, the patient has unresponsive GvHD after 5 days or progressive acute GvHD after 72 hours. If single organ acute GvHD grade II from gut or liver, either progression from single organ or addition of one or two more organs; e.g., if the patient has grade II acute GvHD of the skin, GvHD is more intense and more widespread, or GvHD also includes liver and/or gut.

iv. Patients with steroid refractory GvHD fulfilling the requirements mentioned in a) - c) may be treated with second line therapy, e.g., MMF, serotherapy, ECP, change of CsA for tacrolimus or vice versa, etc. Failure to respond to additional treatment similar to what is described for steroids in c) is necessary before enrolment in this study.

v. Termination of all GvHD medications other than cyclosporine/tacrolimus/MMF and prednisolone is strongly encouraged.

Exclusion criteria

1. Patients with poor performance, not expected to survive 5 days.
2. Patients with a history of hypersensitivity to penicillin and/or gentamycine
3. Poor compliance.

Donor inclusion criteria:

1. MSC donor must be HIV, HB-s antigen, anti HBc and anti HCV negative.
2. First choice original HSC donor HLA-identical sibling donor.
3. Second choice mismatched related or unrelated donor (for instance MSC frozen and left over from another patient).
4. Third choice or emergency pre-expanded third party umbilical cord/placenta derived MSC.

Donor exclusion criteria:

1. Donor more than 65 years of age, or unhealthy.
2. Donor who is positive for HIV, hepatitis Bs antigen, HB-s, anti-HBc and anti HCV negative.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-09; Primary Completion 2012-02 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
GVHD re-staging and/or GVHD mortality ,side effects | within the first 30 days (plus or minus 3 days) after MSC transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Igor B Resnick, MD, PhD, DSci, Principal Investigator — Hadassah University Hospital
Locations (1):
- Hadassah University Hospital, Jerusalem, Israel